CLINICAL TRIAL: NCT02032667
Title: Exercise Games and Physical Activity: Does Multi-player Online Play Improve Adherence?
Brief Title: Exercise Games and Physical Activity: Can a Home-based Exergame System Increase Physical Activity?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Ryan Rhodes, Dr. Ryan Rhodes, University of Victoria
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CCS-701723
Record Dates: First submitted 2013-12-29; First posted 2014-01-10 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Physical Activity
Keywords: physical activity; exergames
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-player condition (Experimental): The multi-player condition examines the aspect of online gaming and social interaction with adherence to the exergame.
  Interventions: Behavioral: Multi-player condition
- Single-player condition (No Intervention): This arm will look at whether those who play an exergame by themselves or with a computer generated player have the same adherence and use when compared to a multi-player condition.

INTERVENTIONS:
Behavioral: Multi-player condition — Children in the multi-player condition will be able to play with and compete against other children in real time.
  Arms: Multi-player condition

SUMMARY:
This study will be investigating an innovative and exciting way to increase physical activity in children between the ages of 9 and 12 years old. Families will be provided with a state-of-the-art exercise bike and video game console to have in their homes. The video games will provide a variety of play including racing, puzzle solving, collaborative play, team play and competitive play. We will be comparing whether a 'multi-player' condition has a greater adherence compared to a 'single-player' condition.

DETAILED DESCRIPTION:
1. Aims of the study: In 2005, the number of deaths attributed to cancer surpassed those caused by major cardiovascular diseases as the number one cause of mortality in Canada, and to this date, continues to significantly impact the lives of Canadians. As a response to the societal and individual afflictions from disease, it is imperative that research initiatives become more focused in the area of primary prevention. Reports have shown that at least half of all new cancer cases and deaths worldwide can be prevented. The largest impact on cancer development are lifestyle variables such as physical activity. Reviews and meta-analysis show a strong inverse linear relationship between physical activity and many of the most prevalent forms of cancer including breast, lung, and colon cancer (i.e., the more an individual exercises the less likely they are to develop cancer). Unfortunately, over 80% of the Canadian populace fails to meet these recommendations. To compound the problem of low physical activity prevalence, the largest declines in activity may occur early in life. Obviously, regular life-long physical activity is the desired outcome for lowering the risk of cancer; thus, promotion efforts targeting critical transitions to physical inactivity early in life are paramount. Two such groups are parents and their children, making family-based physical activity initiatives arguably the most important target for disease prevention. Unfortunately, physical activity interventions focused on the family home are limited and have resulted in negligible changes in physical activity for both children and their parents. Improvements are required in terms of the innovations of interventions.

   An area often overlooked when trying to increase physical participation is affective expectations or judgments (expected pleasure and enjoyment). Affective judgments are a central construct - in some form - in many of our popular health behaviour models, yet few interventions have focused on the modification of affective expectations, despite its reliable and robust association with physical activity. One such group of activities with this potential is interactive exercise videogaming (exergames). Exergaming is a relatively unexplored topic but early results and commentary have been very controversial; the topic has generated as many reviews as it has experimental trials. Overall, the emerging evidence suggests that these games can significantly increase energy expenditure similar to moderate intensity physical activities and these can translate into health-related fitness improvements. The research conducted from our group on this topic also shows this finding. Our studies employ exergames within the context of traditional exercise bikes (i.e., exercise bikes that interact with video games) because they demonstrate physical activity in the moderate to vigorous intensity range that results in marked fitness changes. Despite these positive effects, limited research is available to understand adherence to exergames. Further, of the available literature on exergames and exercise adherence, reviews find that the exergame conditions typically report higher adherence than various control conditions but long-term change is negligible or advantages diminish across time. Our research on the topic mirrors these overall conclusions. For example, in our family-based home pilot study of Game-bike, we showed significantly higher enjoyment and use for children in the exergame condition compared to a control bike across six weeks, yet the prominent differences were within the first three weeks and these were sharply declining in the later weeks. Thus, exergaming research that attempts to foster maintenance is needed to demonstrate that the initial high participation rate can be sustained within the context of the family home. This was the key recommendation from recent systematic reviews of exergames and it forms the rationale for the innovation in this proposal.

   Videogames, similar to these initial exergame results, show decline in playing frequency as games become familiar and the novelty wears. One of the most successful forms of videogaming has been the advent of synchronous multi-player online gaming. Games such as Blizzard's World of Warcraft are played online by millions of people. Specifically, videogames can been played with others online. Gamers may form online social clubs (teams, leagues or "guilds") allowing them to play regularly with the same group of people. The social attachments formed by players can be as strong as those held in the "physical" world, contributing to an extremely long maintenance playtime in comparison to ordinary gaming. To our knowledge, exergames with these properties have not been examined with families in the home. Nevertheless, there is an extensive body of research on the effects of social contexts in supporting physical activity adherence behaviour that suggest that people are more likely to sustain their involvement in a physical activity setting if they participate in social, or group-based, settings rather than on their own. In the context of this trial, if Canadian youth are provided with the opportunity to be part of a virtual group (through online synchronous game play), this will likely support their sense of social connectedness in relation to other youth in that condition, a greater degree of enjoyment of the intervention (affective judgements), and thereafter sustain their adherence behaviours.

   Thus, the primary research question: Does an interactive exergame bike augmented by synchronous online social play capability in comparison to 2) an exergame bike condition both within a family home environment result in greater use among children? Hypothesis: Adherence will be higher for the augmented exergame condition in comparison to the standard exergame condition as children receive the opportunity to play with other children online. The effect will not wane over time from the initial measurement period across three months.

   Our secondary outcomes of parents, physical fitness, total volume of physical activity and perceptions of the bikes will also be examined in the trial. Finally, we will also explore whether season (winter/summer), and gender (males/females) affect the use of the bikes.
2. Study Design and Methods Design: Two-arm parallel design single blinded randomized controlled trial. Participants will be randomised to one of two groups 1) exergame-augmented condition; or 2) exergame standard condition for three months duration. Recruitment: Based on our prior studies, participants will be recruited via advertisements placed through home flyers at elementary/middle schools, cub scouts/brownies, recreation centres, health care centres, children's recreation classes, shopping malls and online interest sites.

Inclusion criteria (see below)

Randomisation and blinding: Families will be randomized at a 1:1 ratio to either intervention or control group, stratified by sex using a central computerised system. Participants will be aware of their group allocation, but all assessors will be blinded to treatment allocation. Justification of sample size: Based on our previous research with exergames, 80 families (40 per group) will be recruited to detect a medium effect size (f2 = .25; (38)) in adherence to physical activity (primary outcome) with a type one error of .05, an average correlation of .75 across time for our DV of interest, and a power of .80. Our sample size also considers the main 2 (group) x 2 (parent/child) x 4 (time) repeated measures design using G-Power and a potential 15% attrition rate.

Procedures and Protocol: After interested participants contact the researcher and are determined to be eligible to participate in the study, families will be visited on site for fitness testing and parents will be asked to complete a brief demographics, physical activity, and quality of life questionnaire while children are asked to complete a brief physical activity and quality of life questionnaire. We will employ a certified exercise physiologist to ensure consistency of the testing. The measurement team will be blind to the treatment conditions of the participants. The family will then be randomized into one of the two conditions. In the standard group, participants will play the games against computer-controlled opponents. In the augmented exergames intervention group, participants will play together, and will be able to talk with each other via a voice over IP link. A Facebook page will be developed allowing the publication of game news, and allowing players to communicate about the game, such as arranging play sessions. For security, only children or parents enrolled in the trail will be permitted to play the game online. The game will be available for play during scheduled times, with separate times for children and for adults.

After the initial six week intervention period, families will be given follow-up questionnaires to complete via an online survey tool. In addition to the brief questionnaires at three months, however, all family members will be asked to participate in a brief end-of-trial qualitative interview to evaluate the impact of the intervention. Although quantitative measurement of outcomes will provide insight into the potency of our exergames intervention, a process evaluation (whereby participants are interviewed) is also essential to examine the content fidelity ("what is done") and process fidelity ("how it is done") of program implementation.

Measures: (See below)

Analysis: Missing data will be evaluated for pattern of missingness for each psychosocial variable and behaviour at all time points using the dummy coding procedures. Depending on the outcome of these tests (e.g., missing at random, missing completely at random, etc.) we will initiate the appropriate missing data handling strategy. ITT analyses will also be performed in addition to sensitivity analysis procedures. A 2 (condition) x 3 (time) repeated measures factorial ANOVA on the primary outcome of child adherence to the bikes. A child from each household in the eligibility range will serve for this analysis (chosen through randomization procedures). Post hoc examinations using Tukey follow-up procedures will be utilized if necessary. Cluster analysis/HLM will be used for parent/child collinearity if needed. The qualitative analyses will incorporate the accuracy, thematic analysis, and coding.

Timeline: We expect the recruitment process to be ongoing across the first two years of the study and continuing for an additional 12 months for data analysis and write-up. The study should be achievable from start to finish in three years (i.e., two-funded years).

ELIGIBILITY:
Inclusion Criteria:

* Participants will be children between the ages of 9 and 12 years old from the greater Victoria, B.C. area and Kingston, Ontario region. Children will be included if they participate in physical activity below Canadian recommended guidelines (for children under 60 minutes of activity daily).
* Participants must also pass the physical activity readiness protocol or seek physician clearance before participation.
* The families must also agree to having the exergaming station in an accessible location in their homes for the duration of the trial
* Will need high speed internet

Exclusion Criteria:

* Children outside of the ages of 9 - 12 years
* Children who are active greater than recommended guidelines (more than 60 minutes of daily activity)
* Children with special needs (i.e. autism spectrum disorder, ADHD/ADD)

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | Baseline, 2 weeks, 4 weeks and 6 weeks.
  Physical activity will be measured via the Physical Activity Questionnaire for Children (PAQ-C) and objective data (use of gamebike) from the exergame. The PAQ-C assesses habitual moderate to vigorous physical activity in children and adolescents.

SECONDARY OUTCOMES:
Change in motivation | Time 1 after first assignment of condition, 2 weeks, 4 weeks and 6 weeks
  Motivation for physical activity will be measured using the constructs of the Theory of Planned Behaviour. These items will measure affective attitude, instrumental attitude, injunctive norm, descriptive norm and perceived behavioural control.
Change in health-related quality of life/psychosocial distress | Baseline, 2 weeks, 4 weeks and 6 weeks.
  Children's Quality of Life will be assessed using the 5-item Satisfaction with Life Scale Adapted for Children (SWLS-C).
Change in health-related fitness | Baseline and 6 weeks
  Body composition, aerobic fitness and musculoskeletal fitness will be measured.
Change in parent and family based leisure time physical activity | Baseline and at follow-up (6 weeks)
  Parent and family based LTPA will be measured by the Godin Leisure Time Exercise Questionnaire and the number of times family based physical activity occurs per week will also be assessed.
Change in equipment and home environment | Baseline
  The home environment questionnaire will look at the availability of physical activity equipment in the home for the child.
Change in sedentary behaviour | Baseline and follow up (6 week)
  Sedentary behaviour of the child will be assessed through parental reported behaviour of their child throughout the week
Change in social support | Baseline and follow up (6-weeks)
  A social support questionnaire will be administered to the child to look at whether parents and friends of the child encourage the child to play sports, to be active and to play the exergame.
Change in elicited beliefs | 2 weeks, 4 weeks and 6 weeks
  The elicited beliefs questionnaire will look at the experience of the child throughout the intervention.
Change in program belonging and social connectedness | 2 weeks, 4 weeks and 6 weeks.
  Examining the sense of connection between players during gameplay throughout the intervention.
Gamer-type | Baseline
  This will be a web-based questionnaire looking at the type of elements in the videogame that the child is attracted to.

OTHER OUTCOMES:
Sociodemographic measures | Baseline
  Sociodemographic measures will include age, parental gender, ethnicity, education, employment status of parents/family, household income, height and weight of parent(s), health status of parent(s).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Rhodes, Doctoral, Principal Investigator — University of Victoria; Nicholas Graham, Doctoral, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - University of Victoria, Victoria, British Columbia
  - Queens University, Kingston, Ontario

REFERENCES:
- [Background] Statistics Canada. Table 102-0561 - Leading causes of death, total population, by age group and sex, Canada, annual, CANSIM (database). Journal [serial on the Internet]. 2012 Date: Available from: http://www5.statcan.gc.ca/cansim/pick-choisir?lang=eng&p2=33&id=1020561.
- [Background] Stein CJ, Colditz GA. Modifiable risk factors for cancer. Br J Cancer. 2004 Jan 26;90(2):299-303. doi: 10.1038/sj.bjc.6601509. PMID 14735167
- [Background] Harvard Report on Cancer Prevention. Volume 1: Causes of human cancer. Cancer Causes Control. 1996 Nov;7 Suppl 1:S3-59. doi: 10.1007/BF02352719. No abstract available. PMID 9091058
- [Background] Adami HO, Day NE, Trichopoulos D, Willett WC. Primary and secondary prevention in the reduction of cancer morbidity and mortality. Eur J Cancer. 2001 Oct;37 Suppl 8:S118-27. doi: 10.1016/s0959-8049(01)00262-3. PMID 11602378
- [Background] Monninkhof EM, Elias SG, Vlems FA, van der Tweel I, Schuit AJ, Voskuil DW, van Leeuwen FE; TFPAC. Physical activity and breast cancer: a systematic review. Epidemiology. 2007 Jan;18(1):137-57. doi: 10.1097/01.ede.0000251167.75581.98. PMID 17130685
- [Background] Tardon A, Lee WJ, Delgado-Rodriguez M, Dosemeci M, Albanes D, Hoover R, Blair A. Leisure-time physical activity and lung cancer: a meta-analysis. Cancer Causes Control. 2005 May;16(4):389-97. doi: 10.1007/s10552-004-5026-9. PMID 15953981
- [Background] Harriss DJ, Atkinson G, Batterham A, George K, Cable NT, Reilly T, Haboubi N, Renehan AG; Colorectal Cancer, Lifestyle, Exercise And Research Group. Lifestyle factors and colorectal cancer risk (2): a systematic review and meta-analysis of associations with leisure-time physical activity. Colorectal Dis. 2009 Sep;11(7):689-701. doi: 10.1111/j.1463-1318.2009.01767.x. Epub 2009 Jan 17. PMID 19207713
- [Background] Colley RC, Garriguet D, Janssen I, Craig CL, Clarke J, Tremblay MS. Physical activity of Canadian adults: accelerometer results from the 2007 to 2009 Canadian Health Measures Survey. Health Rep. 2011 Mar;22(1):7-14. PMID 21510585
- [Background] Colley RC, Garriguet D, Janssen I, Craig CL, Clarke J, Tremblay MS. Physical activity of Canadian children and youth: accelerometer results from the 2007 to 2009 Canadian Health Measures Survey. Health Rep. 2011 Mar;22(1):15-23. PMID 21510586
- [Background] Jedwab J. Actively Canadian: Who's the most active of us all? : Association for Canadian Studies; 2005.
- [Background] Statistics Canada. Canadian Community Health Survey 1994-2003. Government of Canada; 2005 [updated 2005; cited 2005 April 13]; Available from: http://www.acs-aec.ca/Polls/Physical%20Activity%20and%20Obesity.pdf.
- [Background] O'Connor TM, Jago R, Baranowski T. Engaging parents to increase youth physical activity a systematic review. Am J Prev Med. 2009 Aug;37(2):141-9. doi: 10.1016/j.amepre.2009.04.020. PMID 19589450
- [Background] Nasuti G, Rhodes RE. Affective judgment and physical activity in youth: review and meta-analyses. Ann Behav Med. 2013 Jun;45(3):357-76. doi: 10.1007/s12160-012-9462-6. PMID 23297073
- [Background] Rhodes RE, Fiala B, Conner M. A review and meta-analysis of affective judgments and physical activity in adult populations. Ann Behav Med. 2009 Dec;38(3):180-204. doi: 10.1007/s12160-009-9147-y. PMID 20082164
- [Background] Barnett A, Cerin E, Baranowski T. Active video games for youth: a systematic review. J Phys Act Health. 2011 Jul;8(5):724-37. doi: 10.1123/jpah.8.5.724. PMID 21734319
- [Background] Biddiss E, Irwin J. Active video games to promote physical activity in children and youth: a systematic review. Arch Pediatr Adolesc Med. 2010 Jul;164(7):664-72. doi: 10.1001/archpediatrics.2010.104. PMID 20603468
- [Background] Peng W, Crouse JC, Lin JH. Using active video games for physical activity promotion: a systematic review of the current state of research. Health Educ Behav. 2013 Apr;40(2):171-92. doi: 10.1177/1090198112444956. Epub 2012 Jul 6. PMID 22773597
- [Background] Mark R, Rhodes RE, Warburton DER, Bredin SSG. Interactive video games and physical activity: A review of literature and future directions. Health and Fitness Journal of Canada. 2008;1:14-24.
- [Background] Baranowski T, Buday R, Thompson DI, Baranowski J. Playing for real: video games and stories for health-related behavior change. Am J Prev Med. 2008 Jan;34(1):74-82. doi: 10.1016/j.amepre.2007.09.027. PMID 18083454
- [Background] Primack BA, Carroll MV, McNamara M, Klem ML, King B, Rich M, Chan CW, Nayak S. Role of video games in improving health-related outcomes: a systematic review. Am J Prev Med. 2012 Jun;42(6):630-8. doi: 10.1016/j.amepre.2012.02.023. PMID 22608382
- [Background] Warburton DE, Bredin SS, Horita LT, Zbogar D, Scott JM, Esch BT, Rhodes RE. The health benefits of interactive video game exercise. Appl Physiol Nutr Metab. 2007 Aug;32(4):655-63. doi: 10.1139/H07-038. PMID 17622279
- [Background] Warburton DE, Sarkany D, Johnson M, Rhodes RE, Whitford W, Esch BT, Scott JM, Wong SC, Bredin SS. Metabolic requirements of interactive video game cycling. Med Sci Sports Exerc. 2009 Apr;41(4):920-6. doi: 10.1249/MSS.0b013e31819012bd. PMID 19276840
- [Background] Mark RS, Rhodes RE. Testing the effectiveness of exercise videogame bikes among families in the home-setting: a pilot study. J Phys Act Health. 2013 Feb;10(2):211-21. doi: 10.1123/jpah.10.2.211. Epub 2012 Jun 12. PMID 22820629
- [Background] R. K. A Theory of Fun for Game Design. Paraglyph Press; 2004.
- [Background] Yee N. The Demographics, Motivations and Derived Experiences of Users of Massively-Multiuser Online Graphical Environments. PRESENCE: Teleoperators and Virtual Environments. 2006;15:309-29.
- [Background] Dishman RK, Buckworth J. Increasing physical activity: a quantitative synthesis. Med Sci Sports Exerc. 1996 Jun;28(6):706-19. doi: 10.1097/00005768-199606000-00010. PMID 8784759
- [Background] Carron AV, Hausenblas HA, Mack D. Social influence and exercise: A meta-analysis. Journal of Sport & Exercise Psychology. 1996;18:1-16.
- [Background] Casiro NS, Rhodes RE, Naylor PJ, McKay HA. Correlates of intergenerational and personal physical activity of parents. Am J Health Behav. 2011 Jan-Feb;35(1):81-91. doi: 10.5993/ajhb.35.1.8. PMID 20950161
- [Background] Rhodes RE, Naylor PJ, McKay HA. Pilot study of a family physical activity planning intervention among parents and their children. J Behav Med. 2010 Apr;33(2):91-100. doi: 10.1007/s10865-009-9237-0. Epub 2009 Nov 24. PMID 19937106
- [Background] Ye Z, Hernandez H, Graham TCN, Fehlings D, Switzer L, Schumann I. Liberi and the Racer Bike: Exergaming Technology for Children with Cerebral Palsy. ASSETS. in press.
- [Background] Hernandez HA, Graham TCN, Fehlings D, Switzer L, Ye Z, Hamza MA, Savery C, Stach T, editors. Design of an exergaming station for children with cerebral palsy. 30th international conference on Human factors in computing systems - CHI '12; 2012; Austin, Texas.
- [Background] Public Health Agency of Canada. Canada's family guide to physical activity (6-9 years of age). Journal [serial on the Internet]. 2002 Date: Available from: http://www.phac-aspc.gc.ca/pau-uap/paguide/child_youth/pdf/kids_family_guide_e.pdf.
- [Background] Canadian Society for Exercise Physiology. Canadian physical activity guidelines. Journal [serial on the Internet]. 2011 Date: Available from: http://www.csep.ca/english/view.asp?x=804
- [Background] Canadian Society for Exercise Physiology. Physical activity readiness questionnaire. Journal [serial on the Internet]. 2012 Date: Available from: http://www.csep.ca/english/view.asp?x=698.
- [Background] Rhodes RE, Warburton DE, Bredin SS. Predicting the effect of interactive video bikes on exercise adherence: An efficacy trial. Psychol Health Med. 2009 Dec;14(6):631-40. doi: 10.1080/13548500903281088. PMID 20183536
- [Background] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Background] Faul F, Erdfelder E. GPOWER: A priori, post hoc, and compromise power analyses for MS DOS. 2.0 ed. Bonn, Germany: Dept. of Psychology; 1992.
- [Background] King AC, Stokols D, Talen E, Brassington GS, Killingsworth R. Theoretical approaches to the promotion of physical activity: forging a transdisciplinary paradigm. Am J Prev Med. 2002 Aug;23(2 Suppl):15-25. doi: 10.1016/s0749-3797(02)00470-1. PMID 12133734
- [Background] Travers KD. The social organization of nutritional inequities. Soc Sci Med. 1996 Aug;43(4):543-53. doi: 10.1016/0277-9536(95)00436-x. PMID 8844955
- [Background] Travers KD. Using qualitative research to understand the socio-cultural origins of diabetes among Cape Breton Mi'kmaq. Chronic Diseases in Canada. 1995;16:140-3.
- [Background] Dumas JE, Lynch AM, Laughlin JE, Phillips Smith E, Prinz RJ. Promoting intervention fidelity. Conceptual issues, methods, and preliminary results from the EARLY ALLIANCE prevention trial. Am J Prev Med. 2001 Jan;20(1 Suppl):38-47. doi: 10.1016/s0749-3797(00)00272-5. PMID 11146259
- [Background] Rhodes RE, Blanchard CM, Benoit C, Levy-Milne R, Naylor PJ, Symons Downs D, Warburton DE. Physical activity and sedentary behavior across 12 months in cohort samples of couples without children, expecting their first child, and expecting their second child. J Behav Med. 2014 Jun;37(3):533-42. doi: 10.1007/s10865-013-9508-7. Epub 2013 Apr 19. PMID 23606310
- [Background] Ajzen I. The theory of planned behavior. Organizational Behavior and Human Decision Processes. 1991;50:179-211.
- [Background] Ajzen I. Constructing a theory of planned behavior questionnaire. Journal [serial on the Internet]. 2006 Date: Available from: http://people.umass.edu/aizen/pdf/tpb.measurement.pdf.
- [Background] Brown SG, Rhodes RE. Relationships among dog ownership and leisure-time walking in Western Canadian adults. Am J Prev Med. 2006 Feb;30(2):131-6. doi: 10.1016/j.amepre.2005.10.007. PMID 16459211
- [Background] Rhodes RE, Plotnikoff RC. Can current physical activity act as a reasonable proxy measure of future physical activity? Evaluating cross-sectional and passive prospective designs with the use of social cognition models. Prev Med. 2005 May;40(5):547-55. doi: 10.1016/j.ypmed.2004.07.016. PMID 15749137
- [Background] Rhodes RE, Macdonald HM, McKay HA. Predicting physical activity intention and behaviour among children in a longitudinal sample. Soc Sci Med. 2006 Jun;62(12):3146-56. doi: 10.1016/j.socscimed.2005.11.051. Epub 2006 Jan 9. PMID 16406632
- [Background] Godin G, Jobin J, Bouillon J. Assessment of leisure time exercise behavior by self-report: a concurrent validity study. Can J Public Health. 1986 Sep-Oct;77(5):359-62. No abstract available. PMID 3791117
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Gadermann AM, Schonert-Reichl KA, Zumbo BD. Investigating Validity evidence of the Satisfaction with Life Scale Adapted for Children. Social Indicators Research: An International and Interdisciplinary Journal for Quality-of-Life Measurement. in press.
- [Background] 54. Allison PD. Missing Data. Thousand Oaks: Sage Publications; 2002.
- [Background] Chuang JH, Hripcsak G, Heitjan DF. Design and analysis of controlled trials in naturally clustered environments: implications for medical informatics. J Am Med Inform Assoc. 2002 May-Jun;9(3):230-8. doi: 10.1197/jamia.m0997. PMID 11971884
- [Background] Patton MQ. Qualitative Evaluation and Research Methods. second ed. Newbury Park, NJ: Sage; 1990.
- [Background] Crabtree BF, Miller WL. Doing Qualitative Research. Newbury Park, CA: Sage; 1992.
- [Background] Nintendo Co. Ltd., from R. Consolidated Sales Transition by Region. Journal [serial on the Internet]. 2012 Date: Available from: http://www.nintendo.co.jp/ir/library/historical_data/pdf/consolidated_sales_e1206.pdf.
- [Background] BBC News. Microsoft Kinect 'fastest-selling device on record'. Journal [serial on the Internet]. 2011 Date: Available from: http://www.bbc.co.uk/news/business-12697975.
- [Background] Entertainment Software Association. Industry Facts. Journal [serial on the Internet]. 2009 Date: Available from: http://www.theesa.com/facts/index.asp.
- [Background] Entertainment Software Association. Essential Facts About the Computer and Video Game Industry. Journal [serial on the Internet]. 2012 Date: Available from: http://www.theesa.com/facts/pdfs/ESA_EF_2012.pdf.
- [Background] New York Times. Exercise games don't make kids more active. Journal [serial on the Internet]. 2012 Date: Available from: http://www.nytimes.com/2012/06/24/business/active-video-games-dont-make-youths-more-active.html?_r=0.
- [Background] Manske SR, editor. Explaining knowledge use among clients of the Program Training & Consultation Centre. Toronto; 2001; University of Toronto.
- [Background] Lee RG, Garvin T. Moving from information transfer to information exchange in health and health care. Soc Sci Med. 2003 Feb;56(3):449-64. doi: 10.1016/s0277-9536(02)00045-x. PMID 12570966
- [Result] Williams D, Ducheneaut N, Li X, Zhang Y, Yee N, Nickell E. From Tree House to Barracks: The Social Life of Guilds in World of Warcraft. Games and Culture. 2006;1:338-61.
- [Derived] Kaos MD, Beauchamp MR, Bursick S, Latimer-Cheung AE, Hernandez H, Warburton DER, Yao C, Ye Z, Graham TCN, Rhodes RE. Efficacy of Online Multi-Player Versus Single-Player Exergames on Adherence Behaviors Among Children: A Nonrandomized Control Trial. Ann Behav Med. 2018 Sep 13;52(10):878-889. doi: 10.1093/abm/kax061. PMID 30212848